CLINICAL TRIAL: NCT05065944
Title: A Prospective Randomized Trial Comparing Pre-Anesthesia Evaluation Remotely Via Telemedicine Versus in Person for Surgical Patients at H. Lee Moffitt Cancer Center
Brief Title: Comparing Pre-Anesthesia Evaluation Via Telemedicine Versus in Person for Surgical Patients at Moffitt Cancer Center
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-21353
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Gynecologic Cancer; Prostate Cancer; Patient Satisfaction
MeSH Terms: conditions — Prostatic Neoplasms; Patient Satisfaction | interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Anesthesia Evaluation: Telemedicine: Pre-Anesthesia evaluation conducted remotely via video conferencing
  Interventions: Behavioral: Telemedicine
- Pre-Anesthesia Evaluation: In person: Pre-Anesthesia evaluation conducted in person
  Interventions: Behavioral: In Person Visit

INTERVENTIONS:
Behavioral: Telemedicine — Pre-anesthesia assessment (history and physical examination) via telemedicine. Intervention is a one-time telemedicine clinic visit for approximately 30 minutes to 1 hour. Individual patients will be randomized to telemedicine and that visit will be scheduled via the Zoom video conferencing platform.
  Groups: Pre-Anesthesia Evaluation: Telemedicine
Behavioral: In Person Visit — Pre-anesthesia assessment (history and physical examination) in person at Moffitt Cancer Center (usual care)
  Groups: Pre-Anesthesia Evaluation: In person

SUMMARY:
This is a randomized controlled trial of patients scheduled for hysterectomy or prostatectomy surgeries who undergo a pre-anesthesia evaluation at Moffitt Cancer Center PreAnesthesia Testing (PAT) clinic. Traditionally, patients who met certain criteria based on type of surgery or comorbidities would undergo an in-person evaluation in our clinic. In order to make our patient's care more convenient and accessible, investigators have introduced telemedicine evaluation for a certain subset of patients meeting specific criteria. Investigators aim with this randomized trial to investigate the hypothesis that telemedicine pre-anesthesia evaluation is non-inferior to in-person evaluation from the standpoint of day of surgery cancellation rate.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English
* Able to provide signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Presurgical patients at Moffitt Cancer Center scheduled to undergo any type of hysterectomy/salpingo-oophorectomy or prostatectomy surgeries.
* Possesses appropriate equipment (i.e., computer, tablet, smartphone) to undergo telemedicine evaluation.

Exclusion Criteria:

* Patients with documented or observable significant cognitive barriers, hearing, or speech impairment. Examples include a patient who is not alert or oriented, who is unable to sign his or her own surgical consent due to cognitive issues or who cannot understand and repeat back to study coordinator reason for study. If these barriers will not be an issue for a video phone call and can be reasonably accommodated, we will do so. However, our telemedicine technology is still very basic, and these patients may be more comfortable communicating with providers and expressing their needs during an in-person visit
* Surgery 3 days or less away from clinic visit. As in-person assessment is the gold standard, we need to allow some time in case a patient cannot work the technology for a telemedicine visit or an issue comes up where visit needs to be converted to in-person.
* Out of state patients as there are currently medical licensing concerns with conducting telemedicine on patients physically located out of state during the visit.
* Determined to be ineligible for surgery during evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients scheduled for hysterectomy/salpingo-oophorectomy or prostatectomy at Moffit Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients that elect to participate | Up to day 26
  Acceptability of pre-anesthesia telemedicine evaluation will be measured as ≥ 50% of eligible patients consent to participate and ≥ 70% submit exit survey.
Percentage of participants satisfied with telemedicine visit | Up to day 26
  Acceptability will be measured as ≥ 70% strongly agreeing or agreeing with the statement that they were satisfied with their telemedicine visit on an exit survey.

SECONDARY OUTCOMES:
Evaluation of pre-anesthesia evaluation via telemedicine vs in-person | Up to day 30
  Efficacy of pre-anesthesia evaluation via telemedicine will be determined by day of surgery and 48 hours before surgery cancellation rate (number of cancelled appointments divided by number of scheduled appointments).

CONTACTS AND LOCATIONS:
Overall Officials: Nasrin N Aldawoodi, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/clinical-trials/?gclid=EAIaIQobChMImIymzIa-9gIVAZ2GCh3uzAWJEAAYASAAEgI0ovD_BwE